CLINICAL TRIAL: NCT03419208
Title: Randomized Controlled Trial of the Scleroderma Patient-centered Intervention Network Hand Exercise Program
Brief Title: Scleroderma Patient-centered Intervention Network (SPIN) Hand Program
Acronym: SPIN-HAND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Davis Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); The Arthritis Society, Canada (Other)
Responsible Party: Principal Investigator, Brett D Thombs, Professor, Faculty of Medicine, McGill University Senior Investigator, Lady Davis Institute for Medical Research, Jewish General Hospital, Lady Davis Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 12-123A
Record Dates: First submitted 2018-01-26; First posted 2018-02-01 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Scleroderma; Systemic Sclerosis
Keywords: Systemic Sclerosis; Scleroderma; Hand Function; Intervention; Exercise; Telerehabilitation; eHealth; Physical Therapy
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPIN-HAND Program (Experimental): Offered the SPIN-HAND program
  Interventions: Other: SPIN-HAND Program
- Treatment as usual (No Intervention): Not offered SPIN-HAND program, treatment as usual

INTERVENTIONS:
Other: SPIN-HAND Program — The internet-based SPIN-HAND program consists of 4 modules (1) Thumb Flexibility and Strength (3 exercises); (2) Finger Bending (3 exercises); (3) Finger Extension (3 exercises); and (4) Wrist Flexibility and Strength (2 exercises). The program includes sections on developing a personalized program, goal-setting strategies and examples, progress tracking, sharing goals and progress with friends and family, and patient stories of experiences with hand disability and hand exercises. Instructional videos demonstrate and explain how to perform each exercise properly with pictures to illustrate common mistakes. Separate versions of each exercise are available for patients with mild/moderate and more severe hand involvement.
  Arms: SPIN-HAND Program

SUMMARY:
The Scleroderma Patient-centered Intervention Network (SPIN) is an organization established by researchers, health care providers, and people living with scleroderma (systemic sclerosis or SSc) from Canada, the USA, and Europe. The objectives of SPIN are (1) to assemble a large cohort of SSc patients to complete outcome assessments regularly in order to learn more about important problems faced by people living with SSc and (2) to develop and test a series of internet-based interventions to help patients manage aspects of their disease, including hand limitations.

In SSc, approximately 90% of patients experience significant hand function limitations, which impact overall disability more than any other aspect of the disease. The SPIN hand exercise program was designed by SPIN experts in rehabilitation, behavioural therapies, and e-health interventions, as well as patient representatives in SPIN. The program core consists of 4 modules that address specific aspects of hand function, and integrates tools to support key components of successful self-management programs, including goal-setting and feedback, social modeling, and mastery experiences.

The SPIN-HAND trial is a pragmatic randomized control trial (RCT) embedded in the SPIN Cohort that will evaluate the effect of SPIN's online hand exercise program, in addition to usual care, on hand function and health related quality of life (HRQL) in SSc patients with at least mild hand function limitations. SPIN will randomize 586 SPIN Cohort participants with at least mild hand function limitations and an indicated interest in using an online hand exercise program to be offered the hand exercise program or usual care only.

DETAILED DESCRIPTION:
For individuals with SSc, skin and tendon involvement of the hands with significant functional impairment is nearly universal. Hand function limitations impact disability more than any other aspect of the disease. However, given the challenges of conducting high-quality, adequately powered clinical trials and disseminating disease management tools in a rare disease context, proven rehabilitation interventions, including those for hands, are typically not available to rare disease patients. To address this gap, the Scleroderma Patient-centered Intervention Network (SPIN) was founded to (1) assemble a large, multinational cohort of SSc patients as a framework for large-scale rehabilitation and self-management intervention trials; and (2) to develop, test, and disseminate effective disease management tools to patients with SSc.

The SPIN Cohort currently includes over 2000 English- and French-speaking patients from over 40 sites in Canada, the USA, France, and the United Kingdom. SPIN Cohort patients complete outcome measures via the internet upon enrolment and subsequently every 3 months. SPIN utilizes the cohort multiple RCT (cmRCT) design as a framework for conducting trials of interventions. SPIN Cohort patients consent to allow their data to be used for observational research, to assess intervention trial eligibility and, if eligible, be randomized. They also consent that if eligible and randomized to usual care, their data can be used to evaluate intervention effectiveness without them being notified that they have been randomized to the usual care group and not offered the intervention. Thus, in SPIN trials, trial status is masked for patients in the control arm, but not the intervention arm.

The SPIN-HAND trial will evaluate the effect on hand function and HRQL of offering SPIN's online hand exercise program, in addition to usual care, to Cohort patients who have at least mild hand function limitations. The SPIN hand exercise program was designed by SPIN experts in rehabilitation, behavioural therapies, and e-health interventions, as well as patient representatives in SPIN. The program core consists of 4 modules that address specific aspects of hand function, including (1) Thumb Flexibility and Strength (3 exercises); (2) Finger Bending (3 exercises); (3) Finger Extension (3 exercises); and (4) Wrist Flexibility and Strength (2 exercises). The program also integrates tools to support key components of successful self-management programs, including goal-setting and feedback, social modeling, and mastery experiences. 586 SPIN Cohort participants will be enrolled in SPIN-HAND. Eligible patients will be able to use the online intervention in English or French, have at least mild hand function limitations (Cochin Hand Function Scale (CHFS) ≥ 3) and have indicated high interest in using an online hand exercise intervention (≥6 on 0-10 scale).

Randomization will occur at the time of patients' regular SPIN Cohort assessments. Eligible patients, based on questionnaire responses, will be randomized automatically with a 3:2 ratio, using a feature in the SPIN Cohort platform, which provides immediate randomization and complete allocation sequence concealment. A 3:2 ratio is being used in order to increase the number of patients who receive the intervention and to support secondary analyses that examine compliers versus non-compliers.

Trial outcomes will be assessed immediately pre-randomization and at 3 months, 6 months, 12 months, and 24 months post-randomization via the SPIN Cohort for both patients randomized to be offered the intervention and patients who receive usual care only. The primary outcome analysis will compare CHFS scores between eligible patients offered the intervention and those not offered the intervention at 3 months post-randomization. Secondary outcomes will include patient-reported health status, usage logs, user satisfaction, and HRQL.

Statistical analyses will be done blind to trial arm allocation. For the primary analysis, an intent-to-treat approach that compares all patients randomized to be offered versus not offered the intervention will be used. Intervention effects will be estimated using a generalized linear model, adjusted for baseline CHFS scores, recruitment centre, sex, age, disease duration, and diffuse versus limited SSc status. Missing data effects will be investigated using multiple imputation.

Analysis of secondary outcome variables and time points will be done similarly. In addition, complier-average causal effect analysis will be used to estimate effects among patients who accept the intervention offer compared to similar patients in the usual care group. Analysis of usage log data will be conducted to understand the association of uptake and use patterns with intervention effect.

ELIGIBILITY:
Inclusion Criteria:

* SPIN Cohort inclusion criteria:

  1. A SSc diagnosis based on 2013 American College of Rheumatology/European League Against Rheumatism criteria confirmed by a SPIN physician
  2. Be ≥18 years old, be able to give informed consent
  3. Be fluent in English or French.
* For SPIN-HAND:

  1. At least mild hand function limitations (Cochin Hand Function Scale (CHFS) ≥ 3)
  2. Have indicated high interest in using an online hand exercise intervention (≥6 on 0-10 scale) and indicated willingness to participate in a trial of the SPIN-HAND program (yes/no)

Exclusion Criteria:

1. Participants not able to access or respond to questionnaires via the internet are excluded
2. Participants randomized to the intervention group in the SPIN-HAND feasibility study are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Difference in Cochin Hand Function Scale (CHFS) scores between patients offered the intervention and those not offered the intervention 3-months post-randomization | 3 months post-randomization
  The 18-item CHFS measures ability to perform daily hand-related activities (e.g., kitchen, dressing oneself, hygiene, writing/typing). Items are scored on a 0-5 Likert scale (0=without difficulty; 5=impossible). Higher scores indicate less functionality. The total score is obtained by adding the scores of all items (range 0-90).

SECONDARY OUTCOMES:
Difference in Cochin Hand Function Scale (CHFS) scores between patients offered the intervention and those not offered the intervention 6-months post-randomization | 6 months post-randomization
Difference in Cochin Hand Function Scale (CHFS) scores between patients offered the intervention and those not offered the intervention 12-months post-randomization | 12 months post-randomization
Difference in Cochin Hand Function Scale (CHFS) scores between patients offered the intervention and those not offered the intervention 24-months post-randomization | 24 months post-randomization
Difference in Patient Reported Outcomes Measurement Information System (PROMIS-29) profile version 2.0 scores between patients offered the intervention and those not offered the intervention 3-months post-randomization | 3 months post-randomization
  The PROMIS-29 measures 8 domains of health status with 4 items for each of 7 domains (physical function, anxiety, depression, fatigue, sleep disturbance, social roles and activities, pain interference) plus a single item for pain intensity. Items are scored on a 5-point scale (range 1-5), with different response options for different domains, and the single pain intensity item is measured on an 11-point rating scale. Higher scores represent more of the domain being measured; that is, better physical function and ability to participate in social roles and activities, but higher levels of anxiety, depression, fatigue, sleep disturbance, pain interference, and pain intensity.
Difference in Patient Reported Outcomes Measurement Information System (PROMIS-29) profile version 2.0 scores between patients offered the intervention and those not offered the intervention 6-months post-randomization | 6 months post-randomization
Difference in Patient Reported Outcomes Measurement Information System (PROMIS-29) profile version 2.0 scores between patients offered the intervention and those not offered the intervention 12-months post-randomization | 12 months post-randomization
Difference in Patient Reported Outcomes Measurement Information System (PROMIS-29) profile version 2.0 scores between patients offered the intervention and those not offered the intervention 24-months post-randomization | 24 months post-randomization
Difference in European Quality of Life-5 Dimensions (EQ-5D) scores between patients offered the intervention and those not offered the intervention 3-months post-randomization | 3 months post-randomization
  The EQ-5D is a 5-item standardized questionnaire, measuring 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). The items are rated from 1 (no problems) to 3 (extreme problems). Scores range from -0.59 to 1.00 and reflect overall HRQL
Difference in European Quality of Life-5 Dimensions (EQ-5D) scores between patients offered the intervention and those not offered the intervention 6-months post-randomization | 6 months post-randomization
Difference in European Quality of Life-5 Dimensions (EQ-5D) scores between patients offered the intervention and those not offered the intervention 12-months post-randomization | 12 months post-randomization
Difference in European Quality of Life-5 Dimensions (EQ-5D) scores between patients offered the intervention and those not offered the intervention 24-months post-randomization | 24 months post-randomization
Usage log data | Through study completion, 24 months post-randomization
  Device (desktop, tablet, mobile), total time spent on intervention and modules, number of logins, number of times multimedia components are accessed, goal sharing, and use of worksheets
Participant reported satisfaction with the SPIN-HAND exercise program | 3 months post-randomization
  The Client Satisfaction Questionnaire (CSQ-8) is an 8 item questionnaire evaluating user satisfaction. Items are scored on a 4-point Likert scale. Total scores range from 8 to 32, with higher scores indicating higher satisfaction with the service. Items have been modified slightly to refer to the SPIN-HAND program, as opposed to a generic service.

CONTACTS AND LOCATIONS:
Overall Officials: Luc Mouthon, MD, PhD, Principal Investigator — Hôpital Cochin, Paris, France
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Kwakkenbos L, Jewett LR, Baron M, Bartlett SJ, Furst D, Gottesman K, Khanna D, Malcarne VL, Mayes MD, Mouthon L, Poiraudeau S, Sauve M, Nielson WR, Poole JL, Assassi S, Boutron I, Ells C, van den Ende CH, Hudson M, Impens A, Korner A, Leite C, Costa Maia A, Mendelson C, Pope J, Steele RJ, Suarez-Almazor ME, Ahmed S, Coronado-Montoya S, Delisle VC, Gholizadeh S, Jang Y, Levis B, Milette K, Mills SD, Razykov I, Fox RS, Thombs BD. The Scleroderma Patient-centered Intervention Network (SPIN) Cohort: protocol for a cohort multiple randomised controlled trial (cmRCT) design to support trials of psychosocial and rehabilitation interventions in a rare disease context. BMJ Open. 2013 Aug 7;3(8):e003563. doi: 10.1136/bmjopen-2013-003563. PMID 23929922
- [Derived] Kwakkenbos L, Carrier ME, Welling J, Levis B, Levis AW, Sauve M, Turner KA, Tao L, Aguila K, Carboni-Jimenez A, Canedo-Ayala M, Harb S, van den Ende C, Hudson M, van Breda W, Nguyen C, Boutron I, Rannou F, Thombs BD, Mouthon L; SPIN Investigators. Randomized controlled trial of an internet-based self-guided hand exercise program to improve hand function in people with systemic sclerosis: the Scleroderma Patient-centered Intervention Network Hand Exercise Program (SPIN-HAND) trial. Trials. 2022 Dec 12;23(1):994. doi: 10.1186/s13063-022-06923-4. PMID 36510233